CLINICAL TRIAL: NCT02599857
Title: The Effects of a CONCOR Smartphone Application on Arrhythmia, Heart Failure Events and Quality of Life in Patients With Congenital Heart Disease: a Randomized Controlled Trial
Brief Title: The Effects of a CONCOR Smartphone Application
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never started
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Mark Schuuring, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-126481
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2015-11

CONDITIONS: Congenital Heart Disease; Smartphone Application; Arrhythmia; Heart Failure; mHealth; Mobile Health
MeSH Terms: conditions — Heart Defects, Congenital; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONCOR smartphone application (Experimental): Use of CONCOR smartphone application
  Interventions: Device: CONCOR smartphone application
- Standard care (no CONCOR smartphone application) (No Intervention): No CONCOR smartphone application

INTERVENTIONS:
Device: CONCOR smartphone application
  Arms: CONCOR smartphone application

SUMMARY:
Life expectancy of children with congenital heart disease (CHD) has increased dramatically during the past years, due to the successes of cardiac surgery. Nearly all of these children with CHD can be operated at young age and more than 90% reach adulthood. However, many adults with CHD are life-long affected by cardiac events, particularly arrhythmias and heart failure, putting them at risk of premature death. These events have a large impact on quality of life of patients and their families and merit life-long hospital visits in a medical center specialized in adult CHD. Especially for adults with CHD patient care with a smartphone is suited because of their young age and chronic condition. So far, data are lacking on smartphone interventions in patients with CHD.

DETAILED DESCRIPTION:
The investigators aim to determine feasibility of CONCOR smartphone application management in adults with CHD. Moreover, during a twelve months follow up period the investigators aim to evaluate whether management with a CONCOR smartphone application results in a lower rate of heart failure events and arrhythmia as well as a better quality of life than usual care, because of increased patient awareness, behavioral stimuli, healthy life style reminders and more precise medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with CHD being an Academic Medical Center (AMC) patient and/ or patients registered in the Dutch CONCOR registry
* Owning a smartphone

Exclusion Criteria:

* Mental retardation and/ or Down syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Estimated); Primary Completion 2017-05-01 (Estimated); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite of arrhythmia and heart failure events | 1 year

SECONDARY OUTCOMES:
Quality of life questionnaire | 1 year
Mortality | 1 year
Medication adherence questionnaire | 1 year
Usability and learnability questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands